CLINICAL TRIAL: NCT05325788
Title: Developing e-Covery, an App-based Intervention to Support Individuals With Co-occurring Problem Alcohol and Opioid Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2000031915; 1F31AA028992-01 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use Disorder; Opioid Use Disorder
Keywords: intervention development; technology; mHealth; substance use disorder
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single daily message followed by location-based messaging (Other): Participants in this condition receive a single daily message through the intervention app for two weeks (14 days) followed by location-based messaging for two weeks (14 days).
  Interventions: Other: e-Covery; Other: Comparator Condition
- Location-based messaging followed by single daily message (Other): Participants in this condition receive location-based messaging through the intervention app for two weeks (14 days) followed by a single daily message for two weeks (14 days) .
  Interventions: Other: e-Covery; Other: Comparator Condition

INTERVENTIONS:
Other: e-Covery — Through the e-Covery app, participants will receive place-specific messages, sent when participants pass locations identified as triggers.
Other: Comparator Condition — Through the e-Covery app, participants will receive a single general message sent daily in the morning.

SUMMARY:
This project aims to improve the health of individuals engaged in co-occurring alcohol and opioid use by supporting the maintenance of behavior change initiated in substance use treatment. Building on prior research, this study will entail a stage 1b pilot to test the feasibility and acceptability of an app-based intervention for individuals reporting co-occurring alcohol and opioid use. The intervention will involve modifying an app currently used in a research study to collect GPS information to send push notifications when individuals encounter self-identified place-based triggers. Thirty individuals completing substance use treatment will consent to use the app for a thirty-day pilot period and will complete assessments of intervention feasibility and acceptability. Using within-subject tests, the analysis will summarize participant responses to assessments and will compare the use of general messaging to place-specific messaging.

DETAILED DESCRIPTION:
Co-occurring alcohol and opioid use is a public health issue in need of attention and has been linked to various health concerns, such as motor vehicle accidents and drug poisoning and overdose. Individuals engaged in polysubstance use face myriad challenges in sustaining recovery after completion of substance use treatment and return to use after treatment completion is common. One challenge faced by individuals in early recovery is how specific places can serve as triggers for cravings that can precipitate return to use. Smartphone apps have the potential to curtail the effects of such triggers by providing messaging (or "nudging") when individuals are in locations identified as triggers of return to use. To date, research on app-based interventions has yet to examine the effect of such "nudging" independently and has not looked at its effectiveness in addressing co-occurring alcohol and opioid use.

This project aims to improve the health of individuals engaged in co-occurring alcohol and opioid use by supporting the maintenance of behavior change initiated in substance use treatment. Building on prior research, this study will entail a stage 1b pilot to test the feasibility and acceptability of an app-based intervention for individuals reporting co-occurring alcohol and opioid use. The intervention will involve modifying an app currently used in a research study to collect GPS information to send push notifications when individuals encounter self-identified place-based triggers. Thirty individuals completing substance use treatment will consent to use the app for a thirty-day pilot period and will complete assessments of intervention feasibility and acceptability. Using within-subject tests, the analysis will summarize participant responses to assessments and will compare the use of general messaging to place-specific messaging.

ELIGIBILITY:
Inclusion Criteria:

* speak English
* report enrollment in a substance use treatment program at baseline
* report use above the screening tool thresholds for problem alcohol use
* own a smartphone
* reside in Connecticut at baseline with no plans to move in the following month

Exclusion Criteria:

* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the e-Covery app measured by average time spent using the app assessed at day 28 | Day 28
  Feasibility is assessed by average time spent using the app, measured through app usage metrics. More time spent using the app indicates more engagement.
Feasibility of the e-Covery app assessed through qualitative interviews | Day 28
  Feasibility is assessed based on participant responses to questions during an interview taking place after the 28-day pilot period. Participants will be asked about the ease of using the e-Covery app and responses will be coded and analyzed to identify themes related to feasibility. Qualitative findings will be compared to the quantitative findings above using an integrated analysis characteristics of mixed methods approaches.
Average acceptability rating of the e-Covery app measured by 5-point Likert scale | up to Day 28
  Average acceptability is assessed at Days 14 and 28 based on participants' opinion of and satisfaction with the intervention, measured through completion of daily surveys assessing elements of acceptability using Likert scale response options. Higher ratings correspond to higher intervention acceptability. Intent of the outcome measure is to assess the average score from Day 1 through Day 14 compared to the average score from Day 15 through Day 28 to compare the average ratings between conditions.
Acceptability of the e-Covery app assessed through qualitative interviews | Day 28
  Acceptability is assessed based on participant responses to questions during an interview taking place after the 28-day pilot period. Participants will be asked about their satisfaction with the e-Covery app and intervention and responses will be coded and analyzed to identify themes related to acceptability. Qualitative findings will be compared to the quantitative findings above using an integrated analysis characteristics of mixed methods approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Viera, Principal Investigator — Yale University School of Public Health
Locations (1):
- ENRICH Lab, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT05325788/ICF_000.pdf